CLINICAL TRIAL: NCT07170618
Title: A Prospective, Multicenter, Objective Performance Criteria Study to Evaluate the Efficacy and Safety of a Balloon Microcatheter for Clinical Use
Brief Title: Efficacy and Safety of a New Balloon Microcatheter in the Treatment of Intracranial Artery Stenosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sinomed Neurovita Technology Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SINOMED-BMC-2025
Record Dates: First submitted 2025-08-28; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Intracranial Artery Stenosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- balloon microcatheter (Experimental): For the treatment of intracranial artery stenosis, balloon microcatheter would combine the advantages of balloon dilatation first and then, if necessary, the additional deployment of a self-expandable stent via the same balloon microcatheter lumen.
  Interventions: Device: balloon microcatheter

INTERVENTIONS:
Device: balloon microcatheter — The balloon microcatheter simultaneously possesses both balloon dilatation and device delivery functions.

SUMMARY:
The primary objective of this trial is to evaluate the safety and efficacy of a new balloon microcatheter in patients with intracranial artery stenosis.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, objective performance criteria clinical trial to evaluate the safety and efficacy of a balloon microcatheter in the treatment of intracranial artery stenosis. A total of 56 patients are planned to be included. The endpoints include device success, target vessel dissection, target vessel occlusion, mortality and cerebrovascular events, assessed during the in-hospital until discharge.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 80 years of age
2. Patients with intracranial artery stenosis (Degree of stenosis: ≥70%)
3. Target vessel reference diameter must be visually estimated to be 1.25 mm to 4.50 mm
4. Willingness to participate in this clinical trial and signing the consent form for patients or their legally authorised representatives

Exclusion Criteria:

1. The proximal end of the target vessel is extremely tortuous, severely angulated, or heavily calcified, making it difficult for the device to reach the target vessel
2. Pre-existing severe respiratory, hepatic, or renal diseases (e.g., creatinine ≥ 3.0 mg/dL) or coagulation disorders
3. Disabling stroke with a baseline mRS score ≥ 3 points
4. Non-atherosclerosis diseases
5. Patients with stroke caused by branch occlusion
6. Patients who were participating in other clinical trials who had not yet reached the primary clinical endpoint
7. Known hypersensitivity to aspirin, heparin, anesthetics and contrast agents
8. Investigators consider the patient who is not suitable for enrolling in the present trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of device success | During interventional procedure
  The system was successfully delivered to the target site, the balloon was successfully inflated at the lesion area, the therapeutic device was successfully delivered via the microcatheter, and the system was successfully withdrawn.

SECONDARY OUTCOMES:
Incidence of cerebrovascular events, including transient ischemic attack (TIA), ischemic stroke, and hemorrhagic stroke. | Perioperatively (During the in-hospital until discharge)
Rate of target vessel dissection, target vessel occlusion | Perioperatively (During interventional procedure)
  Number of patients with dissection or occlusion of the target vessel
Mortality | Perioperatively (During the in-hospital until discharge)
  The proportion of patients who died during the in-hospital until discharge
Proportion of adverse events or severe adversary event | Perioperatively (During the in-hospital until discharge)
  The proportion of adverse events or severe adverse event
Incidence of device defects | Perioperatively (During the in-hospital until discharge)
  The proportion of device defects in the process of testing, such as label errors, quality problems, malfunctions, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Harbin Medical University, Harbin, China